CLINICAL TRIAL: NCT04596605
Title: Gastrointestinal Tolerance Assessment of T2309
Acronym: GATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT2309-001
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2309 (Experimental): 4 capsules daily for 12 weeks
  Interventions: Other: T2309
- Nutrof Total (Active Comparator): 2 capsules daily for 12 weeks
  Interventions: Dietary Supplement: Nutrof Total

INTERVENTIONS:
Other: T2309 — Food for Special Medical Purpose / 4 capsules daily for 12 weeks
  Arms: T2309
Dietary Supplement: Nutrof Total — 2 capsules daily for 12 weeks
  Other Names: Food Supplement
  Arms: Nutrof Total

SUMMARY:
Gastrointestinal Tolerance assessment of T2309 compared to a food supplement in 50 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Volunteer with no history of gastrointestinal disorders
* Volunteer agreeing not to consume a food supplement other than IP during the study period
* Registered, or agreeing to be registered, in the National Registry of Healthy Volunteers

Exclusion Criteria:

* Any known or suspected hypersensitivity or allergy
* History of or active severe chronic disease or relevant systemic condition incompatible with the study
* Pregnancy or breast-feeding or have planned pregnancy in the next 4 months
* Childbearing potential woman neither surgically sterilized nor using an adequate contraception
* Inability of the subject to understand the study procedures or to give informed consent
* Non-compliant subject
* Participation in this study at the same time as another clinical investigation/study
* Subject having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros
* Subject being institutionalized because of legal or regulatory order, inmate of psychiatric wards, prison or state institutions, or employee of the study site or of the Sponsor's company
* Subject not covered by the government health care scheme of the country in which he/she is living
* Subject with previous, current or anticipated prohibited treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance assessment | 12-week
  Change from baseline in the mean of the daily composite score of gastrointestinal tolerance assessed with the Bristol Stool Scale (BSS) (composite score of stool frequency and consistency) and 10-point Likert scales filled (sum of the ratings of the 4 gastrointestinal symptoms scores) daily for 1 week prior to the completion of the 12-week treatment period (expressed in arbitrary unit/day (a.u./day), range 0-50)

SECONDARY OUTCOMES:
Composite score of gastrointestinal tolerance | 6 weeks
  Change from baseline in the mean of the daily composite score of gastrointestinal tolerance assessed with the BSS and 10-point Likert scales filled daily for 1 week prior to the completion of the 6-week treatment period (a.u./day, range 0-50)
Each component of the composite score of gastrointestinal tolerance | 6 weeks and 12 weeks
  Change from baseline in the mean of each component of the composite score of gastrointestinal tolerance after 6 weeks and 12 weeks of treatment: 4 gastrointestinal symptoms (a.u./day, range 0-10), stool frequency (number of stools/day), stool consistency (a.u./stool, range 1-7)
Acceptability | 6 weeks and 12 weeks
  Assessed by a self-questionnaire to measure the global satisfaction (4-point scales)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Investigation Clinique, Nantes, France

IPD SHARING:
Plan to Share IPD: No